CLINICAL TRIAL: NCT04074642
Title: OCT-angiography as a Pronostic Marker for Visual Impairment in Patients Undergoing Neurosurgery for Compressive Macroadenoma : a Prospective Study.
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-AOI-06
Record Dates: First submitted 2019-08-20; First posted 2019-08-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-03

CONDITIONS: Pituitary Adenoma
Keywords: macroadenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Neurosurgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non compressive adenoma (No Intervention): Optical Coherence Tomography Angiography without surgery
- Compressive adenoma (Experimental): Optical Coherence Tomography Angiography before and after neurosurgery
  Interventions: Procedure: Neurosurgery

INTERVENTIONS:
Procedure: Neurosurgery — adenoma removal
  Arms: Compressive adenoma

SUMMARY:
The aim of the study is to assess accurancy of OCT angiography as a pronostic marker for patients undergoing neurosurgery for compressiver macroadenoma as compared with visual acuity, visual field and OCT.

ELIGIBILITY:
Inclusion Criteria:

* pituitary compressive adenoma (for experimental group)
* pituitary non compressive adenoma

Exclusion Criteria:

* retinian disease
* amblyopia
* parkinson disease
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
change of middle deviation | before surgery (= inclusion), 4 months after surgery and 10 months after surgery
  visual field evolution assessed by Middle deviation
Change of visual function index | before surgery (= inclusion), 4 months after surgery and 10 months after surgery
  visual field evolution assessed by visual function index

CONTACTS AND LOCATIONS:
Overall Officials: ARNAUD MARTEL, Principal Investigator — ophtalmology department, Nice University Hospital
Locations (2):
- France (2):
  - CHU de NICE, Nice
  - Hôpital Pasteur 2 - Service d'Ophtalmologie, Nice